CLINICAL TRIAL: NCT02213536
Title: Investigating the Efficacy of Scalp Sparing Radiotherapy Treatment to the Whole Brain: Examining the Effect of Hair Loss and Re-growth
Brief Title: Investigating the Efficacy of Hair Sparing Radiotherapy Treatment to the Whole Brain.
Acronym: SPARE
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment and follow up
Sponsor: HCA International Limited (Other)
Responsible Party: Principal Investigator, Lynsey RICE, Research and Development radiographer, HCA International Limited
Other Study IDs: HCA
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Brain Cancer
Keywords: Metastatic brain cancer; Whole brain radiotherapy; Scalp sparing whole brain radiotherapy; Prophylactic whole brain radiotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy; Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VMAT WBRT: Patients requiring whole brain radiotherapy as part of their cancer managment.
  Interventions: Radiation: VMAT (Volumetric Modulated Arc Therapy)

INTERVENTIONS:
Radiation: VMAT (Volumetric Modulated Arc Therapy) — Delivering a prescribed radiation dose to the whole brain using VMAT to reduce dose to hair follicles on scalp.
  Other Names: Radiation Therapy; Radiation Oncology

SUMMARY:
To investigate the use of a scalp sparing technique of radiotherapy treatment designed to treat the whole brain. Current treatment methods to treat the whole brain with radiotherapy result in complete alopecia as a side effect. Hair loss is usually patchy and uneven and re-growth similar and slow.

It is hoped that reducing the radiation dose to the hair bearing follicle on the scalp will reduce hair loss and increase the speed and evenness of re-growth.

DETAILED DESCRIPTION:
Rationale for conducting the SPARE study:

The purpose of this study is to evaluate the effect of delivering WBRT via the VMAT method on hair loss and subsequent re-growth. Hair loss has been found to have a negative impact on QoL and can be particularly stressful for patients with a very short life expectancy, this is already well documented. Trying to minimise this treatment side effect, as previously stated in the literature, is a worthwhile investigation. This study is not looking at any prescribed dose changes to the established, evidence based and well documented prescriptions for WBRT. SPARE is an observational study of hair loss and re-growth during and after a patient's prescribed clinical treatment.

Aims and Objectives;

1) To observe hair loss and re-growth in patients undergoing Whole Brain Radiotherapy using the Volumetric Modulated Arc Therapy method of delivery.

As complete alopecia is expected in 100% of patients receiving conventionally delivered WBRT it will be considered a positive result if complete hair loss does not happen when using VMAT in this group of patients.

Assessment of hair loss and re-growth.

The assessment of hair loss and subsequent re-growth will be conducted using both objective and subjective assessments:

1. Objective assessment: Photographic
2. Subjective assessment: Patient interviews \ completion of a hair record sheet.

Photographic assessment:

Initial baseline photographs will be taken before any radiotherapy treatment is delivered on day one of the treatment schedule. Four photographs in total of the head, two laterals (left and right sides), the top (superior) and back (posterior). Subsequent serial photographs will be taken at two weeks, one, two, three, and four months after radiotherapy treatment.

Subjective assessment:

Patients will be asked to give their own opinion on their hair loss \ gain and this will be recorded on the hair record forms and completed by a member of the study team. This will be conducted at the same time intervals as the scalp photographs being taken.

Scalp photos will also be assessed by 2 independent members of the research team and scored using the same scales as the participant. Subsequent follow-up scalp pictures will be assessed against baseline (day 1) photos or complete alopecia images to assess re-growth.

Planning and Dosimetry:

Treatment plans will be generated using a 2 arc VMAT technique generated on Varian's Eclipse treatment planning system using 10 MV photons delivered on a Varian Clinac equipped with a Millennium Multileaf Collimator. Plans will be optimized selecting a maximum dose rate of 600 MU/min.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18
* Positive cancer diagnosis
* Either proven brain metastasis or prophylaxis for primary lung cancer
* Have no epilating chemotherapy planned
* Basic understanding of English

Exclusion Criteria:

* Previous whole brain radiotherapy
* Pregnant females
* Unable to give informed consent
* Urgent cases that need same or next day treatment when referred

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a positive cancer diagnosis requiring whole brain radiotherapy with a life expectancy greater than 4 months.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
To assess hair loss and hair regrowth in patients undergoing WBRT using VMAT via photographic assessment by independent professionals at intervals up to 16 weeks post end of treatment. | 4 months post radiotherapy treatment

SECONDARY OUTCOMES:
To assess patient perceptions of hair loss and hair regrowth in patients undergoing WBRT using VMAT via self assessment at intervals up to 16 weeks post end of treatment. | 4 months post radiotherapy treatment end

CONTACTS AND LOCATIONS:
Overall Officials: David Landau, DR, Study Chair — Clinical Oncologist with practising privilages at The Harley Street Clinic, HCA International Limited hospitals.
Locations (1):
- The Harley Street Clinic, London, United Kingdom